CLINICAL TRIAL: NCT02620267
Title: Target Engagement of the Early Auditory Processing Network by Transcranial Direct Current Stimulation (tDCS): A Pilot Study
Brief Title: Target Engagement of the Early Auditory Processing Network by Transcranial Direct Current Stimulation (tDCS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Walter Dunn, MIRECC Research Fellow, VA Greater Los Angeles Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2015-050587
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia
Keywords: Mismatch Negativity; Transcranial Direct Current Stimulation; MMN; tDCS
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tDCS Stimulation (Experimental): Each subject will receive all three types of stimulation on separate days- anodal, cathodal, and sham stimulation
  Interventions: Device: tDCS Stimulation

INTERVENTIONS:
Device: tDCS Stimulation — Subjects will receive tDCS stimulation over the auditory cortex for 20 min. For anodal stimulation the anode electrodes will be placed over the auditory cortex. For cathodal stimulation, the cathode electrodes will be placed over the auditory cortex. For sham stimulation, the anode electrodes will be placed over the auditory cortex and current turned on for 30 sec before being turned off to simulate the sensation of active stimulation.

SUMMARY:
Individuals with schizophrenia have difficulties in functioning in the community. No one really knows what factors determine how well patients manage in the real world. The purpose of this pilot study is to try a new approach to improving a potential determinant of good community functioning, namely how we process sounds. Specifically, we propose to examine the benefit of transcranial direct current stimulation (tDCS), a new tool that is being developed as a safe and non-invasive neurostimulation method, for improving processing of sounds. Transcranial direct current stimulation involves placing a wet sponge electrode on the head and one on the arm. Electrical current from a device powered by a 9-volt battery will flow from one electrode to the other. A small portion of the current will pass through the skull and stimulate the brain. This procedure is non-invasive and painless and it results in increase or decrease of spontaneous neuronal firing in the brain. Neurons are brain cells that send electrochemical messages to each other. Its safety and beneficial effect on mental functions has been demonstrated in healthy individuals and several clinical populations.

The purpose of this study is to determine if transcranial direct current stimulation can effect how we process sounds.

DETAILED DESCRIPTION:
Neurocognitive and social cognitive deficits are increasingly recognized as core features of schizophrenia. The severity of these deficits closely correlate to functional impairment and patient outcomes in this population. Current pharmacological treatments do not address these illness domains and psychosocial interventions that do are not consistently available. Underlying these higher level cognitive domains are basic sensory processing deficits in the auditory and visual realm that contribute to higher order dysfunction. Evidence of these sensory defects are not readily apparent on clinical exam and are best appreciated using functional imaging and electrophysiological measures. Interventions that remediate these sensory deficits may lead to functional improvement as sensory level improvements may cascade up to higher cognitive domains.

Deficits in auditory processing are evidenced using EEG based event related potentials (ERP). A robust measure of early auditory processing deficits in schizophrenia is the use of an auditory oddball paradigm to elicit Mismatch Negativity (MMN). The MMN ERP is generated when a rare deviant signal is detected in the context of a series of standards. The amplitude of the MMN in schizophrenia patients is decreased compared to healthy controls which reflects a deficit in detecting novel stimuli. This decreased auditory MMN has been shown to be closely correlated with deficits in auditory emotion recognition tasks in subjects with schizophrenia and patient functional outcomes.

This deficit in early auditory processing is thought to be secondary to regions of cortical hypoactivity. Transcranial direct current stimulation (tDCS) is a non-invasive neuromodulation technique that targets cortical regions with direct current and can either increase or decrease cortical excitability depending on the polarity of the tDCS electrode. The MMN network is composed of several generators that serve to process the auditory signal, establish an auditory memory trace, and signal the appearance of the deviant signal. The initial aim of this proposed study will be to determine if tDCS stimulation over the auditory cortex can modulate early auditory processing as measured by the MMN response. Our second aim will be to determine the effect of tDCS stimulation over the auditory cortex on performance measures of auditory processing as assessed by a tone matching task.

Aims and Hypotheses

Aim 1 Determine whether the early auditory processing network can be engaged and modulated by tDCS of the superior temporal lobe, where the earliest generators of the network maybe located, as assessed by changes in the auditory mismatch negativity ERP.

Hypothesis 1 Active tDCS stimulation of the superior temporal lobe will modulate the early auditory processing network resulting in an effect measurable by amplitude changes in the mismatch negativity ERP compared to control sham stimulation.

Aim 2 Determine the effect of tDCS at the temporal generators on the early auditory processing network as assessed by the tone matching task performance measure

Hypothesis 2 Active tDCS stimulation of the temporal generators will modulate the early auditory processing network resulting in a performance change on the tone-matching task compared to sham control stimulation.

Study Protocol

The study will be a within subject, cross over design counterbalanced for order of both stimulation condition and post-stimulation measurement. All patients will receive anodal, cathodal and sham stimulation targeted bilaterally to the superior temporal region (unipolarity, dual-site stimulation). We do not have a directional prediction for the active stimulations (anode and cathode) in terms of increasing or decreasing the amplitude of the MMN ERP, but we do expect active stimulation to change the MMN ERP amplitude. Patients with schizophrenia will be randomly assigned to one of six block stimulation sequences counterbalanced for order of stimulation condition. The goal will be to have complete and usable data from 12 subjects, and thus up to 30 subjects will be enrolled to account for screen failures and drop-outs. At the first visit, subjects will be screened, assessed, and consented if they meet selection criteria. They will then be randomized to one of the counterbalanced stimulation sequences and receive their first stimulation session followed by EEG assessment and tone matching task. Subjects will return in one week for visit 2 and the following week for visit 3. At visits 2 and 3, subjects will receive a tDCS session followed by EEG and tone matching task assessment. All visits will be separated by at least 1 week to washout the effect from the previous stimulation. Each patient will return for a total of 3 stimulation visits.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-V diagnosis of Schizophrenia
2. Estimated premorbid IQ > 70 (based on WRAT reading ability)
3. Understand spoken English sufficiently to comprehend testing procedures
4. Clinically stable: no psychiatric inpatient hospitalization in the last three months, no significant changes in their antipsychotic medications during the previous 6 weeks, and no significant changes in their living situation in the last two months based on data from the registry and self-report
5. Ability to provide signed informed consent and cooperate with study procedures

Exclusion Criteria:

1. No metal in the cranium, intracardiac lines, cardiac pacemaker, medication pump, or increased intracranial pressure
2. No clinically significant neurological or other medical disease as determined by medical history (e.g., seizure disorder, stroke, heart disease, degenerative disease)
3. No history of serious head injury (e.g., loss of consciousness more than 1 hour)
4. No physical, cognitive, or language impairment of such severity as to adversely affect the validity of data
5. No evidence moderate or severe drug or alcohol use disorder in the past six months, and not intoxicated at time of testing
6. No pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Mismatch Negativity- Auditory Oddball Paradigm | 20 min after each stimulation condition

SECONDARY OUTCOMES:
Tone Matching Task | 40 min after each stimulation condition
  Performance based measure of tone discrimination